CLINICAL TRIAL: NCT06839963
Title: Validation of the Kinshasa Lung Ultrasound Approach for the Narrowing of Differential Diagnosis in Children Admitted With Acute Respiratory Symptoms in Low-resource Settings
Brief Title: Kinshasa Lung Ultrasound Approach Validation
Acronym: K-LUS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: HCR24007
Record Dates: First submitted 2025-01-30; First posted 2025-02-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Disease; Children, Only
Keywords: acute respiratory symptoms; children
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study team will perform a prospective, observational study in two sites in the Democratic Republic of Congo (DRC) and Bangladesh in children aged 3 months to 14 years, admitted to hospital with acute respiratory symptoms. The Kinshasa lung ultrasound (K-LUS) approach integrates existing WHO clinical guidelines, lung ultrasound diagnostic accuracy evidence and paediatric ultrasound guidelines. The approach was built using a modified Delphi technique and integrates six LUS profiles, two clinical history features (timing of onset, trauma) and one clinical examination feature (fever) to suggest one among 10 clinical diagnosis. After the initial diagnosis is established by the treating physician, a research assistant will perform a LUS examination and apply the K-LUS approach. Comparison between the K-LUS derived diagnosis and the clinical diagnosis will be performed. After patient discharge a panel will also establish the most likely diagnosis according to all information available during patient stay.

This study is funded by the Wellcome Trust (ITPA grant) ref: WT-ITPA 2021/001

DETAILED DESCRIPTION:
Acute respiratory distress represents one of the main reasons for hospital admission in low and middle income countries. Prompt and accurate diagnosis of the underlying pathological process is crucial to guide appropriate management. Lung Ultrasound (LUS) is an innovative, non-invasive, low-cost, point-of-care tool with high diagnostic accuracy for acute pulmonary diseases. It is a superior alternative to chest radiography (CXR), which is costly and seldom available in low-resource hospitals. To date, we lack a validated LUS-enhanced paediatric diagnostic approach specifically designed for low-resource settings. The primary objective is to test whether a paediatric diagnostic algorithm integrating key elements of patient history, the presence of fever and a systematic bedside LUS examination, changes the admission diagnosis. We also seek to describe the frequency of predefined suspected diagnoses observed and semiquantify pulmonary aeration in children admitted with respiratory symptoms. We will perform a prospective, two-center observational study in the Democratic Republic of Congo (DRC) and Bangladesh in children aged 3 months to 14 years, admitted to hospital with acute respiratory symptoms and signs. The 'Kinshasa lung ultrasound' diagnostic approach (K-LUS) was developed by a group of paediatric clinical and imaging experts based on existing WHO clinical guidelines, published LUS evidence-based frameworks, primary LUS literature on single pathologies and existing paediatric point of care ultrasound guidelines. After the initial diagnosis is established by the treating physician, a research assistant will perform a LUS examination and apply the K-LUS approach, to observe whether there is a change in the initial diagnosis. This is a purely observational study and no intervention will be applied, neither will the patient treatment be changed in relation to the study. The integration of LUS in the diagnostic approach of the critically ill paediatric patient has the potential of improving outcomes and appropriateness of care. It could provide earlier and low-cost diagnosis in both district and referral hospitals, with a potential expansion to peripheral healthcare facilities and integration in existing integrated management of childhood illness (IMCI) guidelines. Such an approach would also help allocate scarce resources by limiting second line radiological imaging techniques only to patients in need.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 months and 14 years;
* Admitted to the emergency department or ward with cough or difficulty in breathing;

Exclusion Criteria:

* Expected short stay in the emergency department (< 6h)
* Emergency transfer to other facilities
* Refusal of informed consent by attending parent or caregiver, as appropriate
* Lung ultrasound not feasible (e.g. non-availability of a trained physician)

Ages: 3 Months to 14 Years | Sex: All
Age Groups: Child
Study Population: Infants and children aged 3 months old to 14 years old presenting with cough or difficulty in breathing.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
The percentage of diagnostic changes | Immediately after the procedure (K-LUS diagnosis)
  The percentage of diagnostic changes prompted by the K-LUS approach compared with the initial clinical diagnosis given by the treating physician.

SECONDARY OUTCOMES:
Percentage agreement for 10 prespecified WHO clinical diagnoses | Immediately after the procedure (K-LUS diagnosis)
  Percentage agreement for 10 prespecified WHO clinical diagnoses, namely (i) Asthma; (ii) Malaria; (iii) Anaemia/metabolic; (iv) Pneumothorax; (v) Congestive heart failure; (vi) Bronchiolitis; (vii) Pulmonary tuberculosis; (viii) Pneumonia; (ix) Pleural effusion (simple or empyema); (x) Haemothorax.

OTHER OUTCOMES:
The net reclassification index | Immediately after the procedure (K-LUS diagnosis)
  The net reclassification index for parenchymal versus non-parencymal diagnosis prompted by the K-LUS protocol compared with the final diagnosis given by a panel after discharge.
Lung ultrasound score | One time as early as possible after the initial clinical diagnosis (maximum 12 hours after the initial clinical diagnosis)
  An ultrasound clip from each individual zone will be saved to the machine for assessment and scoring and quality control purposes. All lung regions will be scored using the LUS aeration score(11,23).
  * 'A-pattern' defined as horizontal repetitions of the pleural line (A-lines) and scored as '0'.
  * 'B-patterns' scored as '1' when more than two well-spaced B-lines are present that cover less than 50% of the pleural line, or as '2' when B-lines cover more than 50% of the pleural line.
  * 'Consolidation-pattern' will be defined as an anatomical image of consolidation >1 cm in diameter and that will be scored as '3'.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Pisani, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit Faculty of Tropical Medicine, Mahidol University Thailand
Locations (3):
- Chittagong Medical College Hospital, Chittagong, Bangladesh
- Kinshasa School of Public Health, University of Kinshasa, Kinshasa, Democratic Republic of the Congo
- Pujehun Govt Hospital Medical, Pujehun, Sierra Leone

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, data from this study may be shared in a de-identified form with other groups or researchers in accordance with the MORU Data Sharing Policy (http://www.tropmedres.ac/data-sharing-policy).
Supporting Information: Study Protocol, ICF
Access Criteria: Refer to MORU data sharing policy with other researchers to use in the future. https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs

REFERENCES:
- [Background] Pocket Book of Hospital Care for Children: Guidelines for the Management of Common Childhood Illnesses. 2nd edition. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK154447/ PMID 24006557
- [Background] Khemani RG, Smith LS, Zimmerman JJ, Erickson S; Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: definition, incidence, and epidemiology: proceedings from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5 Suppl 1):S23-40. doi: 10.1097/PCC.0000000000000432. PMID 26035358
- [Background] Parvathaneni K, Belani S, Leung D, Newth CJ, Khemani RG. Evaluating the Performance of the Pediatric Acute Lung Injury Consensus Conference Definition of Acute Respiratory Distress Syndrome. Pediatr Crit Care Med. 2017 Jan;18(1):17-25. doi: 10.1097/PCC.0000000000000945. PMID 27673384
- [Background] Ord HL, Griksaitis MJ. Fifteen-minute consultation: Using point of care ultrasound to assess children with respiratory failure. Arch Dis Child Educ Pract Ed. 2019 Feb;104(1):2-10. doi: 10.1136/archdischild-2017-313795. Epub 2018 May 25. PMID 29802097
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Singh Y, Tissot C, Fraga MV, Yousef N, Cortes RG, Lopez J, Sanchez-de-Toledo J, Brierley J, Colunga JM, Raffaj D, Da Cruz E, Durand P, Kenderessy P, Lang HJ, Nishisaki A, Kneyber MC, Tissieres P, Conlon TW, De Luca D. International evidence-based guidelines on Point of Care Ultrasound (POCUS) for critically ill neonates and children issued by the POCUS Working Group of the European Society of Paediatric and Neonatal Intensive Care (ESPNIC). Crit Care. 2020 Feb 24;24(1):65. doi: 10.1186/s13054-020-2787-9. PMID 32093763
- [Background] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Background] Marin JR, Abo AM, Arroyo AC, Doniger SJ, Fischer JW, Rempell R, Gary B, Holmes JF, Kessler DO, Lam SH, Levine MC, Levy JA, Murray A, Ng L, Noble VE, Ramirez-Schrempp D, Riley DC, Saul T, Shah V, Sivitz AB, Tay ET, Teng D, Chaudoin L, Tsung JW, Vieira RL, Vitberg YM, Lewiss RE. Pediatric emergency medicine point-of-care ultrasound: summary of the evidence. Crit Ultrasound J. 2016 Dec;8(1):16. doi: 10.1186/s13089-016-0049-5. Epub 2016 Nov 3. PMID 27812885
- [Background] Pereda MA, Chavez MA, Hooper-Miele CC, Gilman RH, Steinhoff MC, Ellington LE, Gross M, Price C, Tielsch JM, Checkley W. Lung ultrasound for the diagnosis of pneumonia in children: a meta-analysis. Pediatrics. 2015 Apr;135(4):714-22. doi: 10.1542/peds.2014-2833. Epub 2015 Mar 16. PMID 25780071
- [Background] Ho MC, Ker CR, Hsu JH, Wu JR, Dai ZK, Chen IC. Usefulness of lung ultrasound in the diagnosis of community-acquired pneumonia in children. Pediatr Neonatol. 2015 Feb;56(1):40-5. doi: 10.1016/j.pedneo.2014.03.007. Epub 2014 Jul 15. PMID 25034957
- [Background] Riviello ED, Kiviri W, Twagirumugabe T, Mueller A, Banner-Goodspeed VM, Officer L, Novack V, Mutumwinka M, Talmor DS, Fowler RA. Hospital Incidence and Outcomes of the Acute Respiratory Distress Syndrome Using the Kigali Modification of the Berlin Definition. Am J Respir Crit Care Med. 2016 Jan 1;193(1):52-9. doi: 10.1164/rccm.201503-0584OC. PMID 26352116
- [Background] Agricola E, Bove T, Oppizzi M, Marino G, Zangrillo A, Margonato A, Picano E. "Ultrasound comet-tail images": a marker of pulmonary edema: a comparative study with wedge pressure and extravascular lung water. Chest. 2005 May;127(5):1690-5. doi: 10.1378/chest.127.5.1690. PMID 15888847
- [Background] Reali F, Sferrazza Papa GF, Carlucci P, Fracasso P, Di Marco F, Mandelli M, Soldi S, Riva E, Centanni S. Can lung ultrasound replace chest radiography for the diagnosis of pneumonia in hospitalized children? Respiration. 2014;88(2):112-5. doi: 10.1159/000362692. Epub 2014 Jul 2. PMID 24992951
- [Background] Papanagnou D, Secko M, Gullett J, Stone M, Zehtabchi S. Clinician-Performed Bedside Ultrasound in Improving Diagnostic Accuracy in Patients Presenting to the ED with Acute Dyspnea. West J Emerg Med. 2017 Apr;18(3):382-389. doi: 10.5811/westjem.2017.1.31223. Epub 2017 Mar 3. PMID 28435488
- [Background] Zanobetti M, Scorpiniti M, Gigli C, Nazerian P, Vanni S, Innocenti F, Stefanone VT, Savinelli C, Coppa A, Bigiarini S, Caldi F, Tassinari I, Conti A, Grifoni S, Pini R. Point-of-Care Ultrasonography for Evaluation of Acute Dyspnea in the ED. Chest. 2017 Jun;151(6):1295-1301. doi: 10.1016/j.chest.2017.02.003. Epub 2017 Feb 16. PMID 28212836
- [Background] Kruisselbrink R, Chan V, Cibinel GA, Abrahamson S, Goffi A. I-AIM (Indication, Acquisition, Interpretation, Medical Decision-making) Framework for Point of Care Lung Ultrasound. Anesthesiology. 2017 Sep;127(3):568-582. doi: 10.1097/ALN.0000000000001779. No abstract available. PMID 28742530
- [Background] Lenahan JL, Volpicelli G, Lamorte A, Jehan F, Bassat Q, Ginsburg AS. Multicentre pilot study evaluation of lung ultrasound for the management of paediatric pneumonia in low-resource settings: a study protocol. BMJ Open Respir Res. 2018 Dec 19;5(1):e000340. doi: 10.1136/bmjresp-2018-000340. eCollection 2018. PMID 30622716
- [Background] Heller T, Wallrauch C, Goblirsch S, Brunetti E. Focused assessment with sonography for HIV-associated tuberculosis (FASH): a short protocol and a pictorial review. Crit Ultrasound J. 2012 Nov 21;4(1):21. doi: 10.1186/2036-7902-4-21. PMID 23171481
- [Background] Snelling PJ, Shefrin AE, Moake MM, Bergmann KR, Constantine E, Deanehan JK, Dessie AS, Elkhunovich MA, Gold DL, Kornblith AE, Lin-Martore M, Nti B, Pade KH, Parri N, Sivitz A, Lam SHF. Establishing the international research priorities for pediatric emergency medicine point-of-care ultrasound: A modified Delphi study. Acad Emerg Med. 2022 Nov;29(11):1338-1346. doi: 10.1111/acem.14588. Epub 2022 Sep 13. PMID 36043227
- [Background] Shefrin AE, Warkentine F, Constantine E, Toney A, Uya A, Doniger SJ, Sivitz AB, Horowitz R, Kessler D. Consensus Core Point-of-care Ultrasound Applications for Pediatric Emergency Medicine Training. AEM Educ Train. 2019 Mar 14;3(3):251-258. doi: 10.1002/aet2.10332. eCollection 2019 Jul. PMID 31360818
- [Background] Ali N, Shakeel E, Soomar SM. Need of Point of Care Ultrasound Training in Pediatric Emergency Medicine Practice: A Wake-Up Call for the Low-Income Countries. Glob Pediatr Health. 2023 Jul 18;10:2333794X231187485. doi: 10.1177/2333794X231187485. eCollection 2023. PMID 37484605
- [Background] Vercesi V, Pisani L, van Tongeren PSI, Lagrand WK, Leopold SJ, Huson MMA, Henwood PC, Walden A, Smit M, Riviello ED, Pelosi P, Dondorp AM, Schultz MJ; Lung Ultrasound Consortium. External confirmation and exploration of the Kigali modification for diagnosing moderate or severe ARDS. Intensive Care Med. 2018 Apr;44(4):523-524. doi: 10.1007/s00134-018-5048-5. Epub 2018 Jan 24. No abstract available. PMID 29368056
- [Background] Pivetta E, Goffi A, Lupia E, Tizzani M, Porrino G, Ferreri E, Volpicelli G, Balzaretti P, Banderali A, Iacobucci A, Locatelli S, Casoli G, Stone MB, Maule MM, Baldi I, Merletti F, Cibinel GA, Baron P, Battista S, Buonafede G, Busso V, Conterno A, Del Rizzo P, Ferrera P, Pecetto PF, Moiraghi C, Morello F, Steri F, Ciccone G, Calasso C, Caserta MA, Civita M, Condo' C, D'Alessandro V, Del Colle S, Ferrero S, Griot G, Laurita E, Lazzero A, Lo Curto F, Michelazzo M, Nicosia V, Palmari N, Ricchiardi A, Rolfo A, Rostagno R, Bar F, Boero E, Frascisco M, Micossi I, Mussa A, Stefanone V, Agricola R, Cordero G, Corradi F, Runzo C, Soragna A, Sciullo D, Vercillo D, Allione A, Artana N, Corsini F, Dutto L, Lauria G, Morgillo T, Tartaglino B, Bergandi D, Cassetta I, Masera C, Garrone M, Ghiselli G, Ausiello L, Barutta L, Bernardi E, Bono A, Forno D, Lamorte A, Lison D, Lorenzati B, Maggio E, Masi I, Maggiorotto M, Novelli G, Panero F, Perotto M, Ravazzoli M, Saglio E, Soardo F, Tizzani A, Tizzani P, Tullio M, Ulla M, Romagnoli E; SIMEU Group for Lung Ultrasound in the Emergency Department in Piedmont. Lung Ultrasound-Implemented Diagnosis of Acute Decompensated Heart Failure in the ED: A SIMEU Multicenter Study. Chest. 2015 Jul;148(1):202-210. doi: 10.1378/chest.14-2608. PMID 25654562
- [Background] Pencina MJ, D'Agostino RB Sr, D'Agostino RB Jr, Vasan RS. Evaluating the added predictive ability of a new marker: from area under the ROC curve to reclassification and beyond. Stat Med. 2008 Jan 30;27(2):157-72; discussion 207-12. doi: 10.1002/sim.2929. PMID 17569110
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558